CLINICAL TRIAL: NCT03945591
Title: A Phase II Study of High-Dose Post-Transplant Cyclophosphamide and Bortezomib (CyBor) for the Prevention of Graft-versus-Host Disease Following Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Brief Title: High-Dose Post-Transplant Cyclophosphamide and Bortezomib (CyBor) for the Prevention of Graft-versus-Host Disease Following Allogeneic Hematopoietic Stem Cell Transplantation (HSCT)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-01185
Record Dates: First submitted 2019-05-08; First posted 2019-05-10 (Actual); Results first posted 2023-12-06 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: GVHD
Keywords: Cyclophosphamide; Bortezomib
MeSH Terms: interventions — Bortezomib; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cyclophosphamide and Bortezomib (Experimental)
  Interventions: Drug: Bortezomib; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Bortezomib — 1.3 mg/m2 IV 6 hours after graft infusion and 72 hours thereafter.
Drug: Cyclophosphamide — 50 mg/kg IV over 2 hours on Day +3 and +4

SUMMARY:
This is a single arm open label phase II clinical trial. Adult patients with hematological malignancies undergoing allogeneic HSCT from matched-related or unrelated donor are eligible for the study if they meet the standard criteria defined in the investigator's institutional standard operation procedures (SOPs), meet all inclusion criteria, and do not satisfy any exclusion criteria. Patients will receive reduced-intensity or myeloablative conditioning regimen of fludarabine, busulfan, and rabbit anti-thymocyte globulin (rATG). Patients will receive PTCyBor as GvHD prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* Karnofsky score ≥ 70%
* No evidence of progressive bacterial, viral, or fungal infection
* Creatinine clearance > 50 mL/min/1.72m2
* Total bilirubin, ALT and AST < 2 x the upper limit of normal (except for Gilbert's syndrome)
* Alkaline phosphatase ≤ 250 IU/L
* Left Ventricular Ejection Fraction (LVEF) > 45%
* Adjusted Carbon Monoxide Diffusing Capacity (DLCO) > 60%
* Negative HIV serology
* Negative pregnancy test: confirmation per negative serum β-human chorionic gonadotropin (β-hCG)

Exclusion Criteria:

* Pregnant or nursing females or women of reproductive capability who are unwilling to completely abstain from heterosexual sex or practice 2 effective methods of contraception from the first dose of bortezomib through 90 days after the last dose. A woman of reproductive capability is one who has not undergone a hysterectomy (removal of the womb), has not had both ovaries removed, or has not been post-menopausal (stopped menstrual periods) for more than 24 months in a row.
* Male subjects who refuse to practice effective barrier contraception during the entire study treatment period and through a minimum of 90 days after the last dose of study drug, or completely abstain from heterosexual intercourse. This must be done even if they are surgically sterilized (i.e., post-vasectomy).
* Inability to provide informed consent.
* Patient had myocardial infarction within 6 months prior to enrollment or has New York Heart Association (NYHA) Class III or IV heart failure (see Appendix E), uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening must be documented by the investigator as not medically relevant.
* Known allergies to any of the components of the investigational treatment regimen.
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Diagnosed or treated for another malignancy within 3 years of enrollment, with the exception of complete resection of basal cell carcinoma or squamous cell carcinoma, an in-situ malignancy, or low-risk prostate cancer after curative therapy.
* Participation in clinical trials with other investigational agents not included in this trial, within 14 days of the start of this trial and throughout the duration of this trial.
* Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2019-06-20 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2024-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad Al-Homsi, MD, Principal Investigator — New York Langone Medical Center
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).Upon reasonable request is likely the most appropriate as well will report on incidental findings (i.e. infections) that may impact transplant.
Supporting Information: SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Requests should be directed to Ankeeta.Joshi@nyulangone.org To gain access, data requestors will need to sign a data access agreement.

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 23 participants were consented. 2 of these participants did not initiate the study.
Period: Overall Study
Arm/Group | Cyclophosphamide and Bortezomib
Started | 21
Completed | 16
Not Completed | 5
Not completed — Participant not transplanted | 1
Not completed — Change in treatment plan | 3
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cyclophosphamide and Bortezomib
Number analyzed (Participants) | 16
Age, Continuous [Median (Full Range); unit: years] | 63 [22 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 14
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 16
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Experience Acute GvHD
Description: Rate of acute GvHD post-transplant. All participants that received a transplant and received any prophylactic treatment will be included in the analysis.
Time Frame: Day 120 Post-Transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclophosphamide and Bortezomib
Number analyzed (Participants) | 13
percentage of participants | 38.46 [22 to 47]

2. Primary Outcome: Percentage of Participants Who Experience Moderate to Severe Chronic GvHD
Description: Rate of chronic GvHD post-transplant. All participants that received a transplant and received any prophylactic treatment will be included in the analysis.
Time Frame: Day 365 Post-Transplant
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cyclophosphamide and Bortezomib
Number analyzed (Participants) | 11
percentage of participants | 36.36 [22 to 46]

3. Secondary Outcome: Incidence of Primary Graft Failure
Description: Incidence of graft failure will be calculated from date of transplant to failure for all patients who receive a transplant and any prophylactic treatment and from date of completion of prophylactic treatment for all participants that completed treatment. Graft failure is defined as failure to achieve neutrophil engraftment by day 28 post-transplant or lack of donor chimerism > 50% by day 45 post-transplant not due to the underlying malignancy.
Time Frame: Day 45 Post-Transplant
Reporting Status: Not Posted

4. Secondary Outcome: Incidence of Poor Graft Function
Description: Incidence of poor graft function will be calculated from date of transplant to failure for all patients who receive a transplant and any prophylactic treatment and from date of completion of prophylactic treatment for all participants that completed treatment. Poor graft function is defined by at least 2 of the following 3 criteria: Hemoglobin < 8 g/dL, ANC < 0.5 109/L, and platelets < 20 109/L. The cytopenia must be unexplained (such as by disease relapse) and unresponsive to cytokines and must last at least 4 weeks.
Time Frame: Day 30 Post-Transplant
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of Secondary Graft Failure
Description: Incidence of secondary graft failure is evaluated after engraftment is achieved; this outcome is calculated from date of engraftment for all patients with engraftment. Secondary graft failure is defined as poor graft function associated with donor chimerism < 5%.
Time Frame: Day 730 Post-Transplant
Reporting Status: Not Posted

6. Secondary Outcome: Treatment Related Mortality (TRM)
Description: Number of participant deaths not attributable to disease relapse or progression . This outcome is analyzed based on participants that who received a transplant with any prophylactic treatment and for all patients who received a transplant and completed prophylactic treatment.
Time Frame: Day 730 Post-Transplant
Reporting Status: Not Posted

7. Secondary Outcome: Relapse Rate (RR)
Description: Percentage of participants in whom the disease for which transplant is performed is evident by methods of disease detection after transplant. This outcome is analyzed for all patients who received a transplant and for all transplanted patients that completed treatment.
Time Frame: Day 730 Post-Transplant
Reporting Status: Not Posted

8. Secondary Outcome: Graft Versus Host Disease Relapse Free Survival (GRFS)
Description: Percentage of participants who are without reported GvHD III-IV acute GvHD, chronic GvHD requiring systemic therapy and have not experienced relapse or death after transplant.
Time Frame: Day 730 Post-Transplant
Reporting Status: Not Posted

9. Secondary Outcome: Overall Survival (OS)
Description: Percentage of participants alive at the end of the study's evaluation period.
Time Frame: Day 730 Post-Transplant
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: From the start of the conditioning regimen for a minimum of 30 days after the last treatment dose (41 days total).
Description: Investigator assessment at each study visit.
Arm/Group | Cyclophosphamide and Bortezomib
All-Cause Mortality (participants affected / at risk) | 1/16
Serious Adverse Events (participants affected / at risk) | 7/16
Other Adverse Events (participants affected / at risk) | 10/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide and Bortezomib (N=16)
Abdominal Pain (Gastrointestinal disorders) | 3
Anemia (Blood and lymphatic system disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Blood Bilirubin Increased (Investigations) | 2
Confusion (Psychiatric disorders) | 1
Cytomegalovirus Infection Reactivation (Infections and infestations) | 3
Death (General disorders) | 1
Fall (Injury, poisoning and procedural complications) | 2
Fever (General disorders) | 4
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypotension (Vascular disorders) | 2
COVID Infection (Infections and infestations) | 3
BK Viremia (Infections and infestations) | 1
Adenovirus (Infections and infestations) | 1
Methemoglobinemia (Blood and lymphatic system disorders) | 1
Sepsis (Infections and infestations) | 1
Syncope (Nervous system disorders) | 4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cyclophosphamide and Bortezomib (N=16)
Agitation (Psychiatric disorders) | 1
Alanine Aminotransferase Increased (Investigations) | 2
Alkaline Phosphatase Increased (Investigations) | 1
Aspartate Aminotransferase Increased (Investigations) | 2
Atrial Fibrillation (Cardiac disorders) | 1
Bacteremia (Infections and infestations) | 1
Bloating (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dizziness (Nervous system disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Epstein-Barr virus infection reactivation (Infections and infestations) | 1
Febrile Neutropenia (Blood and lymphatic system disorders) | 1
Gastric Hemorrhage (Gastrointestinal disorders) | 1
Headache (Nervous system disorders) | 2
Hematuria (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Hypoxia (Infections and infestations) | 1
C. Difficile (Infections and infestations) | 1
Mucositis Oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Pain (General disorders) | 1
Platelet Count Decreased (Investigations) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Secretions (Respiratory, thoracic and mediastinal disorders) | 1
Sinus Tachycardia (Cardiac disorders) | 1
Skin Ulceration (Skin and subcutaneous tissue disorders) | 1
Sore Throat (Respiratory, thoracic and mediastinal disorders) | 1
Upper Gastrointestinal Hemorrhage (Gastrointestinal disorders) | 1
Urinary Tract Infection (Infections and infestations) | 3
Viremia (Infections and infestations) | 3
Vomiting (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/91/NCT03945591/Prot_SAP_000.pdf